CLINICAL TRIAL: NCT03591601
Title: Effectiveness of a Global Manual Therapy Protocol vs Exercises With Foam Rolling for Tension Headache
Brief Title: Effectiveness of Manual Therapy vs Exercises With Foam Rolling for Tension Headache
Acronym: MTvsFR-TTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: ID0021
Record Dates: First submitted 2018-06-01; First posted 2018-07-19 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Tension-type Headache
Keywords: Tension-type headache; Pain
MeSH Terms: conditions — Tension-Type Headache; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual therapy protocol (Active Comparator): Treatment based on manual therapy with proven evidence.
  Interventions: Other: Manual Therapy protocol
- Foam Rolling protocol (Experimental): Treatment based on massage with a Foam Rolling
  Interventions: Other: Foam Rolling protocol
- Placebo Control (Placebo Comparator): Placebo treatment based on the placement of the hands on the head without intention to treat.
  Interventions: Other: Placebo control

INTERVENTIONS:
Other: Manual Therapy protocol — Treatment based on manual therapy with proven evidence.
  Arms: Manual therapy protocol
Other: Foam Rolling protocol — Treatment based on massage with a Foam Rolling
  Arms: Foam Rolling protocol
Other: Placebo control — Placebo treatment based on the placement of the hands on the head without intention to treat.
  Arms: Placebo Control

SUMMARY:
Tension headache (CT) is the most frequent problem within the group of headaches, with a prevalence of 30-78% of the population throughout its life. Regarding this pathology, treatment with manual therapy has been studied a lot, observing the benefits of different techniques separately in elements such as disability, impact or depression.

The "Foam Rolling" (FR) is an element widely used in sport that has been studied its applications in terms of hip and knee flexibility after application in muscles such as the quadriceps or hamstrings.

In this study the investigators recruited randomized subjects in three groups, one of exercises with RF, another of a protocol of manual therapy (TM) techniques and one control (CTR) with a placebo treatment. There will be 4 treatments, 1 per week, and the data will be collected in 3 moments, pre-treatment, post-treatment and one month after treatment.

The investigators will evaluate aspects such as the average pain of headaches, the impact, disability, quality of life, self-satisfaction and pain at the pressure of painful points of the trapezius and suboccipital muscles.

DETAILED DESCRIPTION:
Introduction Primary headaches occupy an important field in neurology consultations. Both migraines and tension headaches are often self-treated by the patients themselves and for some patients, headache is a true disease, constituting a symptomatology that can have various etiologies, from severe to functional organics. Headache, when it becomes chronic, becomes a serious problem for the patient with important repercussions on their quality of life.

Objective. To evaluate the effectiveness of the application of the treatment by means of manual therapy in patients with tension headache and to compare it with the application of massage by means of a roll of foam manufactured for this purpose.

Methodology The study will be carried out in the Faculty of Physiotherapy of the Universitat de València. An experimental, longitudinal and prospective design, controlled, randomized, with 3 groups will be carried out.

Population. The sample will be formed by participants diagnosed with tension headache, following the criteria established by the IHS.

Subjects with headache less than 15 days per month and other types of primary headache, as well as those associated with drug abuse and those who do not meet the criteria established by the IHS, will be excluded from the study.

Experimental treatment The patients will be randomly assigned to 3 different groups (one group of treatment with manual therapy, one group that will receive massage and another group of placebo control).

The treatment will last for 8 weeks (4 weeks of treatment and 4 weeks of follow-up). The 2 groups will be evaluated before treatment, at the end of this and in the follow-up (30 days after treatment).

Evaluations

For the collection of data, a clinical interview with data referring to headache was designed and the following evaluation instruments are included:

* Scale disability due to HDI Headache
* Impact of pain HIT-6
* Quality of life SF-36
* Visual Analog Scale (EVA)
* Algometry. Measurement of pain at pressure on spinous and transverse processes
* CROM. Cervical range
* QS. Body satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 55 years old.
* CT medical diagnosis.
* Evolution of, at least, 3 months of the CT.
* Suffer, at least, 1 crisis a week.
* Meet, at least, 2 of the following IHS criteria:
* Bilateral location.
* Pressure pain, not pulsating pain.
* Having a mild-moderate pain intensity.
* Pain that is not aggravated by physical activity.
* Minimum duration of 30 'of the TC.
* Accompanied by some associated symptom:

or Photophobia. or Fonofobia. or mild nausea.

Exclusion Criteria:

* Have less than 20 years or more than 55.
* Cervical trauma.
* Musculoskeletal problems that may be aggravated by movement.
* Klein test positive.
* Contraindications to receive manual therapy.
* Musculoskeletal problems that may give another type of headache.
* Problems of dizziness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | 8 weeks
  Visual Analog Scale. The participants are asked to mark the intensity of pain from 1 to 10, with 1 being almost non-existent and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Disability headache | 8 weeks
  Headache Disability Index (HDI). Questionnaire developed by G.P. Jacobson et al. to quantify the impact of disability due to headache in daily life. The objective is to identify the difficulties that the patient experiences due to headaches. It consists of two questions: 1) intensity of pain (mild, moderate and severe), and 2) frequency (once a month, more than 1 and less than 4 times a month, and once a week). In addition, it includes 25 items with two subscales, one emotional (13 items) and another functional (12 items) with three possible answers ("no" 0 points, "sometimes" 2 points, "yes" 4 points). The maximum score is 100 points, with 0 "no disability" and 100 "maximum disability".
Impact of headache | 8 weeks
  Headache Impact Test (HIT-6). Published by Ware et al. To measure the impact of headache. The score is calculated as follows: never (6 points), few times (8 points), sometimes (10 points), very often (11 points) and always (13 points). With a total of 49 or less points is considered "little or no impact", between 50-55 "some impact", between 56-59 "significant impact" and 60 or more "very severe impact".
Pressure pain threshold | 8 weeks
  Algometer. To assess the pain threshold at the pressure of the different muscles, a mechanical pressure algometer (Wagner Instruments FDK 20) will be used. The pressure pain threshold is the minimum pressure that is needed to cause pain or discomfort at a certain point. In obtaining the result, the average of the 3 scores obtained from each point was made. The reliability of this procedure is high in healthy subjects [BCI = 0.91 (95% confidence interval: 0.82-0.97)] 28.31. In patients with TMD, reliability is moderate (ICC = 0.64)
Cervical range movment | 8 weeks
  Goniometry. The range of joint movement of the neck is measured by the use of a goniometer. Flexion, extension, lateral tilt and cervical rotation are assessed. To be able to perform the measurement, the patient is asked to remain in a sitting position keeping his back at 90 degrees and his head in a neutral position. The physiotherapist instructs the patients to perform the previously explained movements, until reaching the maximum range of movement or in the presence of pain. We proceed to evaluate mobility in the 3 planes: sagittal plane, frontal plane and transverse plane. 3 measurements of each movement are made, and the final measurement obtained is the average of each previous result.
Body satisfaction | 8 weeks
  Body satisfaction questionnaire. It contains 10 positive and 10 negative adjectives about the participant's body sensation with alternative answers ranging from 1 = Excellent to 5 = Poor. Each question is scored independently.
Health Status | 8 weeks
  SF-36 questionnaire. It consists of 36 items with the following scales: Physical function (items 3a, 3b, 3c, 3d, 3e, 3f, 3g, 3h, 3i, 3j), Physical role (items 4a, 4b, 4c, 4d), Corporal pain ( items 7, 8), General Health (items 1, 11a, 11b, 11c, 11d), Vitality (items 9a, 9e, 9g, 9i), Social function (items 6, 10), Emotional role (items 5a, 5b, 5c) and Mental Health (items 9b, 9c, 9d, 9f, 9h). Includes an item on the change in the general health status with respect to the previous year (item 2). To calculate the score, we must first homogenize the address of the answers by re-coding the items that require it, so that "the higher the score, the better the health condition", then the calculation of the sum of the items of each scale and, finally, the linear transformation of raw scores on a scale of 0 (worst health status for that dimension) to 100 (the best health status).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Physiotherapy, Valencia
  - Gemma V Espí López, Valencia